CLINICAL TRIAL: NCT01519960
Title: A Phase IIIb Parallel Group, Open Label Study of Pegylated Interferon Alfa-2a Monotherapy (PEG-IFN, Ro 25-8310) Compared to Untreated Control in Children With HBeAg Positive Chronic Hepatitis B
Brief Title: A Study of Pegasys (Peginterferon Alfa-2a) Versus Untreated Control in Children With HBeAg Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YV25718; 2011-002732-70 (EudraCT Number)
Record Dates: First submitted 2011-12-06; First posted 2012-01-27 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (4):
- A Pegasys (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- B Untreated Control (No Intervention)
- C Fibrosis non-randomized (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- Switch (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — Body surface area adapted doses of 45-180 mcg subcutaneously weekly for 48 weeks, Weeks 1- 48
  Arms: A Pegasys; C Fibrosis non-randomized
Drug: peginterferon alfa-2a [Pegasys] — Body surface area adapted doses of 45-180 mcg subcutaneously weekly for 48 weeks, after Week 48 for Group B patients who have not experienced HBeAg seroconversion
  Arms: Switch

SUMMARY:
This parallel group, open label study will evaluate the safety and efficacy of Pegasys (peginterferon alfa-2a) versus untreated control in children (age 3 years to <18 years at baseline) with HBeAg positive chronic hepatitis B. Children without advanced fibrosis and without cirrhosis will be randomized 2:1 to treatment Group A, receiving Pegasys 45-180 mcg subcutaneously weekly for 48 weeks, or to the untreated control Group B. Children with advanced fibrosis will be assigned to treatment group C and receive 48 weeks of treatment with Pegasys. Children in the untreated control Group B who have not experienced seroconversion 48 weeks after randomization may enter the Switch Arm to receive 48 weeks of Pegasys treatment. This offer will be available for 1 year following 48 weeks from randomization. Anticipated time on study treatment is 48 weeks. All subjects will be followed up for 5 years after the end of treatment (A,C,Switch)/principal observation (B) period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 3 years to <18 years of age at baseline
* Positive HBsAg for more than 6 months
* Positive HBeAg and detectable HBV DNA at screening
* A liver biopsy obtained within the past 2 years prior to baseline (and more than 6 months after the end of previous therapy for hepatitis B) to confirm the presence of advanced fibrosis or exclude cirrhosis
* Compensated liver disease (Child-Pugh Class A)
* Elevated serum alanine transferase (ALT)
* Normal thyroid gland function at screening

Exclusion Criteria:

* Subjects with cirrhosis
* Subjects must not have received investigational drugs or licensed treatments with anti-HBV activity within 6 months of baseline. Subjects who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded
* Known hypersensitivity to peginterferon
* Positive test results at screening for hepatitis A, hepatitis C, hepatitis D or HIV infection
* History or evidence of medical condition associated with chronic liver disease other than chronic hepatitis B
* History or evidence of bleeding from esophageal varices
* Decompensated liver disease (e.g. ascites, Child-Pugh Class B or C)
* History of immunologically mediated disease
* Pregnant or lactating females

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (6):
  - Univ of California SF, Benioff Children's Hospital; Pediatrics, Gastro, Hepatology & Nutrition, San Francisco, California
  - Johns Hopkins Hospital - Pediatric Gastroenterology, Baltimore, Maryland
  - Children's Hospital Boston-Harvard Medical School; Division of Gastoenterology, Boston, Massachusetts
  - St. Louis University - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Womens and Childrens Hospital; Department of Gastroenterology, North Adelaide, South Australia
  - Royal Children's Hospital; Department of Gastroenterology, Melbourne, Victoria
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Bulgaria (2):
  - Specialized Hospital for Active Treatment of Pediatrics Diseases; Clinic of Gastroenterology, Sofia
  - University Hospital "St. Marine"; Dept. of Pediatrics, Varna
- China (10):
  - Beijing 302 Hospital; No. 2 Infectious Disease Section, Beijing
  - Beijing You An Hospital; Digestive Dept, Beijing
  - the First Hospital of Jilin University, Changchun
  - Southwest Hospital , Third Military Medical University, Chongqing
  - The Eighth People's Hospital of Guangzhou, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The First Affilliated Hospital of Kunming Medical College, Kunming
  - Xinjiang Uygur Autonomous Region Hospital of Chinese Traditional Medicine, Urumqi (乌鲁木齐)
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- HELIOS Klinikum Wuppertal, Zentrum für Kinder- und Jugendmedizin, Universität Witten-Herdecke, Wuppertal, Germany
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Western Galilee Hospital - Nahariya, Nahariya
- Uni Degli Studi Di Bologna - Policlinica S. Orsola; Inst. Di Malattie Infettive, Bologna, Emilia-Romagna, Italy
- Poland (3):
  - Wojewodzki Szpital Obserwacyjno-Zakazny; Oddział Pediatrii, Chorób Infekcyjnych i Hepatologii, Bydgoszcz
  - Krakowski Szpital Specjalistyczny im Jana Pawła II; Oddział Chorób Infekcyjnych Dzieci, Krakow
  - Wojewodzki Specjalistyczny Szpital im. Dr W.Bieganskiego; Oddział Obserwacyjno-Zakażny dla Dzieci, Lodz
- Russia (4):
  - SFI Sceintific Research institute of nutrition of RAMS, Moscow
  - SI Sceintific children health center RAMS, Moscow
  - FSI Scientific research Institute of children's infections, Saint Petersburg
  - MC Gepatolog, Samara
- Ukraine (2):
  - Kyiv Children's Clinical Infectious Diseases Hospital, Kyiv
  - SI Institute of the pediatrics, obstetrics and gynecology, Kyiv
- United Kingdom (3):
  - Birmingham Children'S Hopsital; Liver Unit, Birmingham
  - Kings College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare Trust, London

REFERENCES:
- [Derived] Wirth S, Zhang H, Hardikar W, Schwarz KB, Sokal E, Yang W, Fan H, Morozov V, Mao Q, Deng H, Huang Y, Yang L, Frey N, Nasmyth-Miller C, Pavlovic V, Wat C. Efficacy and Safety of Peginterferon Alfa-2a (40KD) in Children With Chronic Hepatitis B: The PEG-B-ACTIVE Study. Hepatology. 2018 Nov;68(5):1681-1694. doi: 10.1002/hep.30050. Epub 2018 Oct 8. PMID 29689122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 211 individuals were screened for entry into the study. Of these, there were 161 participants enrolled in the study and included in the main analyses.
Groups:
- Group A: PEG-IFN Monotherapy Without Advanced Fibrosis: Participants without advanced fibrosis were randomized and received PEG-IFN monotherapy for 48 weeks with a 24-week follow-up and an additional 4.5-year extended follow-up. Each dose of 45 to 180 micrograms (mcg) was based on BSA and given as a once-weekly subcutaneous (SC) injection for 48 weeks. BSA-based dosing was as follows: 0.51-0.53 square meters (m^2), 45 mcg; 0.54-0.74 m^2, 65 mcg; 0.75-1.08 m^2, 90 mcg; 1.09-1.51 m^2, 135 mcg; greater than (>) 1.51 m^2, 180 mcg.
- Group B: Untreated Control Without Advanced Fibrosis: Participants without advanced fibrosis were randomized and were evaluated for 48 weeks with a 24-week follow-up and an additional ongoing 4.5-year extended follow-up. As the study is open-label, participants did not receive any investigational or placebo treatment during the 48-week principal observation period (POP). For ethical reasons, participants in Group B had a reduced visit schedule (every 12 weeks) compared to participants in Group A through the end of 24-week follow-up. After completing the POP, the same PEG-IFN regimen administered in Group A was offered to participants in Group B who had not experienced hepatitis B envelope antigen (HBeAg) seroconversion. The offer remained for up to 1 year following the Week 48 visit. From the time a given participant switched to PEG-IFN, he/she was no longer included in Group B.
- Group C: PEG-IFN Monotherapy With Advanced Fibrosis: Participants with advanced fibrosis were allocated (not randomized) to receive PEG-IFN monotherapy for 48 weeks with a 24-week follow-up and an additional 4.5-year extended follow-up. Each dose of 45 to 180 mcg was based on BSA and given as a once-weekly SC injection for 48 weeks. BSA-based dosing was as follows: 0.51-0.53 m^2, 45 mcg; 0.54-0.74 m^2, 65 mcg; 0.75-1.08 m^2, 90 mcg; 1.09-1.51 m^2, 135 mcg; >1.51 m^2, 180 mcg.
Period: Overall Study
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Started | 101 | 50 | 10
Completed Week 48 | 99 | 47 | 10
Completed Follow-Up (FU) Week 12 | 99 | 26 | 10
Completed FU Week 24 | 99 | 15 | 10
Completed FU 5 Year | 75 | 28 | 5
Switch Group | 0 | 33 | 0
Completed | 75 | 28 | 5
Not Completed | 26 | 22 | 5
Not completed — Withdrawal from the study | 26 | 22 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis | Group C: PEG-IFN Monotherapy With Advanced Fibrosis | Total
Number analyzed (Participants) | 101 | 50 | 10 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.41 (4.57) | 11.2 (5.01) | 6.7 (3.27) | 10.55 (4.81)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0
  Children (2-11 years) | 53 | 20 | 9 | 82
  Adolescents (12-17 years) | 48 | 30 | 1 | 79
  Adults (18-64 years) | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 18 | 2 | 57
  Male | 64 | 32 | 8 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBeAg Seroconversion at 24 Weeks After End of Treatment (EOT)/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of hepatitis B envelope antibody (anti-HBe). The percentage of participants with HBeAg seroconversion at 24 weeks after EOT/POP was reported. The 95 percent (%) confidence interval (CI) was calculated by the Pearson-Clopper method. Intent-to-Treat (ITT) Population: All randomized participants regardless of treatment received.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 25.7 (17.56) [17.56 to 35.4] | 6 (1.25) [1.25 to 16.55]
Statistical Analysis 1: Comparison: Group A: PEG-IFN Monotherapy Without Advanced Fibrosis vs Group B: Untreated Control Without Advanced Fibrosis; Analysis stratified by hepatitis B virus (HBV) genotype A versus non-A genotypes and alanine aminotransferase (ALT) less than (<) 5 times (×) upper limit of normal (ULN) versus greater than or equal to (≥) 5 × ULN at Baseline. The OR was calculated using Group B as reference; Test type: Other; p = 0.0043, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.43, 95% CI 2-sided [1.54 to 19.2]
Statistical Analysis 2: Comparison: Group A: PEG-IFN Monotherapy Without Advanced Fibrosis vs Group B: Untreated Control Without Advanced Fibrosis; Test type: Other; p = 0.3732, Breslow-Day

2. Secondary Outcome: Percentage of Participants With Loss of HBeAg at 24 Weeks After EOT/POP in Groups A and B
Description: The percentage of participants with loss of HBeAg at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 25.7 (17.56) [17.56 to 35.4] | 6 (1.25) [1.25 to 16.55]

3. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroconversion at 24 Weeks After EOT/POP in Groups A and B
Description: HBsAg seroconversion was defined as loss of HBsAg and the presence of hepatitis B surface antibody (anti-HBs). The percentage of participants with HBsAg seroconversion at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 7.9 (3.48) [3.48 to 15.01] | 0 (0) [0 to 7.11]

4. Secondary Outcome: Percentage of Participants With Normal ALT at 24 Weeks After EOT/POP in Groups A and B
Description: Normal ALT was defined as ALT less than or equal to (≤) ULN, where each ULN was given by the laboratory at which the sample was analyzed. The percentage of participants with normal ALT at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 51.5 (41.33) [41.33 to 61.55] | 12 (4.53) [4.53 to 24.31]

5. Secondary Outcome: Percentage of Participants With HBV Deoxyribonucleic Acid (DNA) <20,000 International Units Per Milliliter (IU/mL) at 24 Weeks After EOT/POP in Groups A and B
Description: HBV DNA was quantified using polymerase chain reaction (PCR) by Roche Taqman. The percentage of participants with HBV DNA <20,000 IU/mL at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 33.7 (24.56) [24.56 to 43.75] | 4 (0.49) [0.49 to 13.71]

6. Secondary Outcome: Percentage of Participants With HBV DNA <2,000 IU/mL at 24 Weeks After EOT/POP in Groups A and B
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <2,000 IU/mL at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 28.7 (20.15) [20.15 to 38.57] | 2 (0.05) [0.05 to 10.65]

7. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <20,000 IU/mL at 24 Weeks After EOT/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <20,000 IU/mL at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 22.8 (15.02) [15.02 to 32.18] | 4 (0.49) [0.49 to 13.71]

8. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <2,000 IU/mL at 24 Weeks After EOT/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <2,000 IU/mL at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 19.8 (12.54) [12.54 to 28.91] | 2 (0.05) [0.05 to 10.65]

9. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at EOT/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. The percentage of participants with HBeAg seroconversion at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 7.9 (3.48) [3.48 to 15.01] | 6 (1.25) [1.25 to 16.55]

10. Secondary Outcome: Percentage of Participants With Loss of HBeAg at EOT/POP in Groups A and B
Description: The percentage of participants with loss of HBeAg at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 8.9 (4.16) [4.16 to 16.24] | 6 (1.25) [1.25 to 16.55]

11. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at EOT/POP in Groups A and B
Description: HBsAg seroconversion was defined as loss of HBsAg and the presence of anti-HBs. The percentage of participants with HBsAg seroconversion at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 6.9 (2.83) [2.83 to 13.76] | 0 (0) [0 to 7.11]

12. Secondary Outcome: Percentage of Participants With Loss of HBsAg at EOT/POP in Groups A and B
Description: The percentage of participants with loss of HBsAg at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 10.9 (5.56) [5.56 to 18.65] | 0 (0) [0 to 7.11]

13. Secondary Outcome: Percentage of Participants With Normal ALT at EOT/POP in Groups A and B
Description: Normal ALT was defined as ALT ≤ ULN, where each ULN was given by the laboratory at which the sample was analyzed. The percentage of participants with normal ALT at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 18.8 (11.72) [11.72 to 27.81] | 22 (11.53) [11.53 to 35.96]

14. Secondary Outcome: Percentage of Participants With HBV DNA <20,000 IU/mL at EOT/POP in Groups A and B
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <20,000 IU/mL at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 36.6 (27.27) [27.27 to 46.81] | 12 (4.53) [4.53 to 24.31]

15. Secondary Outcome: Percentage of Participants With HBV DNA <2,000 IU/mL at EOT/POP in Groups A and B
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <2,000 IU/mL at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 30.7 (21.9) [21.9 to 40.66] | 2 (0.05) [0.05 to 10.65]

16. Secondary Outcome: Percentage of Participants With HBV DNA Undetectable at EOT/POP in Groups A and B
Description: HBV DNA was quantified using PCR by Roche Taqman. Undetectable HBV DNA was defined as HBV DNA <29 IU/mL. The percentage of participants with HBV DNA undetectable at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 18.8 (11.72) [11.72 to 27.81] | 0 (0) [0 to 7.11]

17. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <20,000 IU/mL at EOT/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <20,000 IU/mL at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 6.9 (2.83) [2.83 to 13.76] | 6 (1.25) [1.25 to 16.55]

18. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <2,000 IU/mL at EOT/POP in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <2,000 IU/mL at EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of participants | 6.9 (2.83) [2.83 to 13.76] | 0 (0) [0 to 7.11]

19. Secondary Outcome: Quantitative Serum ALT Level in Groups A and B
Description: Quantitative ALT at each visit was averaged among all participants and expressed as a factor of the laboratory-specific ULN (for example, 1 × ULN, 2 × ULN, 3 × ULN). ITT Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: If number of participants equals 0, the calculation was not performed because no participants provided data for the visit.
Measure: Mean (Standard Deviation); unit: factor of ULN
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
factor of ULN
  Baseline | 2.779 (2.483) | 2.878 (1.997)
  Week 1: number analyzed (Participants) | 101 | 0
  Week 1 | 3.427 (2.687) |
  Week 2: number analyzed (Participants) | 101 | 0
  Week 2 | 2.846 (1.885) |
  Week 4: number analyzed (Participants) | 101 | 0
  Week 4 | 3.343 (2.455) |
  Week 8: number analyzed (Participants) | 101 | 0
  Week 8 | 3.262 (2.797) |
  Week 12: number analyzed (Participants) | 101 | 0
  Week 12 | 3.189 (3.06) |
  Week 18: number analyzed (Participants) | 101 | 0
  Week 18 | 3.036 (2.389) |
  Week 24 | 2.753 (2.725) | 2.401 (2.638)
  Week 30: number analyzed (Participants) | 101 | 0
  Week 30 | 2.587 (2.128) |
  Week 36 | 2.45 (1.856) | 2.341 (2.204)
  Week 42: number analyzed (Participants) | 101 | 0
  Week 42 | 2.316 (1.429) |
  Week 48 | 2.122 (1.389) | 1.954 (1.371)
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | 1.303 (1.74) |
  FU Week 12: number analyzed (Participants) | 101 | 0
  FU Week 12 | 2.064 (2.027) |
  FU Week 24 | 1.477 (1.625) | 1.7 (1.385)

20. Secondary Outcome: Quantitative HBV DNA Level in Groups A and B
Description: Quantitative HBV DNA at each visit was averaged among all participants and expressed in log10 IU/mL. ITT Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
log10 IU/mL
  Baseline | 8.094 (0.986) | 8.056 (0.987)
  Week 12 | 6.49 (2.009) | 7.909 (1.267)
  Week 24 | 5.966 (2.398) | 7.857 (1.327)
  Week 36 | 5.575 (2.513) | 7.685 (1.608)
  Week 48 | 5.224 (2.701) | 7.551 (1.761)
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | 5.739 (2.935) |
  FU Week 12 | 5.914 (3.065) | 7.214 (2.46)
  FU Week 24 | 5.707 (3.113) | 7.2 (2.506)

21. Secondary Outcome: Change From Baseline in Quantitative HBV DNA Level in Groups A and B
Description: The change in quantitative HBV DNA from Baseline to each visit was averaged among all participants and expressed in log10 IU/mL. ITT Population. All participants were included in the endpoint analysis. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
log10 IU/mL
  Week 12 | -1.588 (1.625) | -0.156 (1.093)
  Week 24 | -2.112 (1.996) | -0.168 (1.214)
  Week 36 | -2.525 (2.148) | -0.359 (1.411)
  Week 48 | -2.877 (2.374) | -0.493 (1.518)
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | -2.34 (2.582) |
  FU Week 12 | -2.164 (2.737) | -0.86 (2.163)
  FU Week 24 | -2.381 (2.778) | -0.587 (2.259)

22. Secondary Outcome: Percentage of Participants With Loss of HBeAg at 24 Weeks After EOT in Group C
Description: The percentage of participants with loss of HBeAg at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population: All participants who received at least one dose of study drug (if assigned) and had at least one post-baseline safety assessment.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

23. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at 24 Weeks After EOT in Group C
Description: HBsAg seroconversion was defined as loss of HBsAg and the presence of anti-HBs. The percentage of participants with HBsAg seroconversion at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 0 (0) [0 to 30.85]

24. Secondary Outcome: Percentage of Participants With Loss of HBsAg at 24 Weeks After EOT in Group C
Description: The percentage of participants with loss of HBsAg at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 0 (0) [0 to 30.85]

25. Secondary Outcome: Percentage of Participants With Normal ALT at 24 Weeks After EOT in Group C
Description: Normal ALT was defined as ALT ≤ ULN, where each ULN was given by the laboratory at which the sample was analyzed. The percentage of participants with normal ALT at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 70 (34.75) [34.75 to 93.33]

26. Secondary Outcome: Percentage of Participants With HBV DNA <20,000 IU/mL at 24 Weeks After EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <20,000 IU/mL at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 70 (34.75) [34.75 to 93.33]

27. Secondary Outcome: Percentage of Participants With HBV DNA <2,000 IU/mL at 24 Weeks After EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <2,000 IU/mL at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 70 (34.75) [34.75 to 93.33]

28. Secondary Outcome: Percentage of Participants With HBV DNA Undetectable at 24 Weeks After EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. Undetectable HBV DNA was defined as HBV DNA <29 IU/mL. The percentage of participants with HBV DNA undetectable at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

29. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <20,000 IU/mL at 24 Weeks After EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <20,000 IU/mL at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

30. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <2,000 IU/mL at 24 Weeks After EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <2,000 IU/mL at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

31. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. The percentage of participants with HBeAg seroconversion at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 20 (2.52) [2.52 to 55.61]

32. Secondary Outcome: Percentage of Participants With Loss of HBeAg at EOT in Group C
Description: The percentage of participants with loss of HBeAg at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 20 (2.52) [2.52 to 55.61]

33. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at EOT in Group C
Description: HBsAg seroconversion was defined as loss of HBsAg and the presence of anti-HBs. The percentage of participants with HBsAg seroconversion at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 0 (0) [0 to 30.85]

34. Secondary Outcome: Percentage of Participants With Loss of HBsAg at EOT in Group C
Description: The percentage of participants with loss of HBsAg at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 0 (0) [0 to 30.85]

35. Secondary Outcome: Percentage of Participants With Normal ALT at EOT in Group C
Description: Normal ALT was defined as ALT ≤ ULN, where each ULN was given by the laboratory at which the sample was analyzed. The percentage of participants with normal ALT at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 40 (12.16) [12.16 to 73.76]

36. Secondary Outcome: Percentage of Participants With HBV DNA <20,000 IU/mL at EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <20,000 IU/mL at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 40 (12.16) [12.16 to 73.76]

37. Secondary Outcome: Percentage of Participants With HBV DNA <2,000 IU/mL at EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with HBV DNA <2,000 IU/mL at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

38. Secondary Outcome: Percentage of Participants With HBV DNA Undetectable at EOT in Group C
Description: HBV DNA was quantified using PCR by Roche Taqman. Undetectable HBV DNA was defined as HBV DNA <29 IU/mL. The percentage of participants with HBV DNA undetectable at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 20 (2.52) [2.52 to 55.61]

39. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <20,000 IU/mL at EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <20,000 IU/mL at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 20 (2.52) [2.52 to 55.61]

40. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <2,000 IU/mL at EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The percentage of participants with combined HBeAg seroconversion and HBV DNA <2,000 IU/mL at EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 20 (2.52) [2.52 to 55.61]

41. Secondary Outcome: Quantitative Serum ALT Level in Group C
Description: Quantitative ALT at each visit was averaged among all participants and expressed as a factor of the laboratory-specific ULN (for example, 1 × ULN, 2 × ULN, 3 × ULN). Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: factor of ULN
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
factor of ULN
  Baseline | 2.804 (1.118)
  Week 1 | 3.117 (1.322)
  Week 2 | 2.896 (1.304)
  Week 4 | 2.444 (1.727)
  Week 8 | 2.703 (2.035)
  Week 12 | 2.793 (1.288)
  Week 18 | 2.215 (1.032)
  Week 24 | 1.887 (1.095)
  Week 30 | 2.22 (1.553)
  Week 36 | 2.172 (1.09)
  Week 42 | 1.593 (0.516)
  Week 48 | 1.645 (1.242)
  FU Week 4 | 1.136 (0.506)
  FU Week 12 | 1.521 (0.755)
  FU Week 24 | 1.549 (1.595)

42. Secondary Outcome: Quantitative HBV DNA Level in Group C
Description: Quantitative HBV DNA at each visit was averaged among all participants and expressed in log10 IU/mL. Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 7.866 (0.977)
  Week 12 | 5.782 (1.771)
  Week 24 | 5.599 (2.386)
  Week 36 | 5.2 (2.451)
  Week 48 | 5.319 (2.747)
  FU Week 4 | 4.604 (2.442)
  FU Week 12 | 4.252 (2.596)
  FU Week 24 | 3.694 (3.127)

43. Secondary Outcome: Change From Baseline in Quantitative HBV DNA Level in Group C
Description: The change in quantitative HBV DNA from Baseline to each visit was averaged among all participants and expressed in log10 IU/mL. Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 IU/mL
  Week 12 | -2.084 (1.1)
  Week 24 | -2.267 (1.595)
  Week 36 | -2.529 (1.879)
  Week 48 | -2.546 (2.14)
  FU Week 4 | -3.262 (2.102)
  FU Week 12 | -3.613 (2.519)
  FU Week 24 | -4.15 (2.904)

44. Secondary Outcome: Estimated Area Under the Concentration-Time Curve (AUC) by BSA Category
Description: AUC was estimated using population pharmacokinetic (PK) modeling. The AUC at steady-state was averaged among participants who received PEG-IFN and reported by BSA category. Categories of BSA-based dosing used in the analysis were as follows: 0.54-0.74 m^2, 65 mcg; 0.75-1.08 m^2, 90 mcg; 1.09-1.51 m^2, 135 mcg; >1.51 m^2, 180 mcg. The estimated AUC was expressed in hours by nanograms per milliliter (h*ng/mL). PK Substudy Population: All participants who consented to participate in the PK substudy. "Number of subjects analyzed" reflects the total combined number of participants who provided evaluable data across all BSA categories. The number of participants who provided evaluable data within each BSA category (n) is shown in the table.
Time Frame: Pre-dose (0 hours) at Baseline and Weeks 4, 8, 12, 24; post-dose (24-48, 72-96, 168 hours) during Weeks 1, 24 (up to 24 weeks overall)
Measure: Mean (Full Range); unit: h*ng/mL
Groups:
- All Groups Combined: All participants enrolled in the study
Arm/Group | All Groups Combined
Number analyzed (Participants) | 161
h*ng/mL
  0.54-0.74 m^2 | 3320 [633 to 5064]
  0.75-1.08 m^2 | 4037 [1897 to 6916]
  1.09-1.51 m^2 | 2765 [1750 to 4392]
  >1.51 m^2 | 3448 [1914 to 5000]

45. Secondary Outcome: Percentage of Participants With >15% Drop in Height Percentile for Age in Groups A and B
Description: The percentage of participants with >15% drop in height percentile for age from Baseline to each visit was reported. Safety Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Weeks 12, 24 (up to 72 weeks overall)
Measure: Number; unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 48
percentage of participants
  Week 12 | 1 | 0
  Week 24 | 5 | 8.5
  Week 36 | 4 | 4.2
  Week 48 | 6.1 | 2.1
  FU Week 12 | 10.9 | 4.2
  FU Week 24 | 12 | 6.7

46. Secondary Outcome: Percentage of Participants With >15% Drop in Weight Percentile for Age in Groups A and B
Description: The percentage of participants with >15% drop in weight percentile for age from Baseline to each visit was reported. Safety Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 48
percentage of participants
  Week 4: number analyzed (Participants) | 101 | 0
  Week 4 | 2 |
  Week 8: number analyzed (Participants) | 101 | 0
  Week 8 | 5 |
  Week 12 | 5.1 | 2.1
  Week 18: number analyzed (Participants) | 101 | 0
  Week 18 | 8.1 |
  Week 24 | 16 | 8.5
  Week 30: number analyzed (Participants) | 101 | 0
  Week 30 | 13.1 |
  Week 36 | 11.3 | 8.3
  Week 42: number analyzed (Participants) | 101 | 0
  Week 42 | 13.1 |
  Week 48 | 12.5 | 8.5
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | 8.1 |
  FU Week 12 | 6.9 | 20.8
  FU Week 24 | 11 | 20

47. Secondary Outcome: Quantitative HBeAg Level in Groups A and B
Description: Quantitative HBeAg at each visit was averaged among all participants and expressed in log10 Paul Ehrlich Institute units per milliliter (PEIU/mL). ITT Population. All participants were included in the endpoint analysis. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 PEIU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
log10 PEIU/mL
  Baseline | 2.736 (0.502) | 2.568 (0.65)
  Week 12 | 2.09 (0.879) | 2.391 (0.878)
  Week 24 | 1.865 (0.956) | 2.36 (0.896)
  Week 36 | 1.604 (0.991) | 2.272 (0.985)
  Week 48 | 1.466 (1.053) | 2.124 (1.091)
  FU Week 24 | 1.537 (1.334) | 2.217 (1.395)

48. Secondary Outcome: Quantitative HBsAg Level in Groups A and B
Description: Quantitative HBsAg at each visit was averaged among all participants and expressed in log10 IU/mL. ITT Population. All participants were included in the endpoint analysis. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
log10 IU/mL
  Baseline | 4.309 (0.687) | 4.383 (0.721)
  Week 12 | 3.844 (1.186) | 4.299 (0.809)
  Week 24 | 3.509 (1.507) | 4.336 (0.732)
  Week 36 | 3.265 (1.661) | 4.272 (0.726)
  Week 48 | 3.078 (1.769) | 4.215 (0.718)
  FU Week 24 | 3.37 (1.63) | 4.394 (0.939)

49. Secondary Outcome: Quantitative HBeAg Level in Group C
Description: Quantitative HBeAg at each visit was averaged among all participants and expressed in log10 PEIU/mL. Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 PEIU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 PEIU/mL
  Baseline | 2.344 (0.981)
  Week 12 | 1.62 (1.288)
  Week 24 | 1.802 (1.14)
  Week 36 | 1.561 (1.178)
  Week 48 | 1.429 (1.259)
  FU Week 24 | 1.442 (1.416)

50. Secondary Outcome: Quantitative HBsAg Level in Group C
Description: Quantitative HBsAg at each visit was averaged among all participants and expressed in log10 IU/mL. Safety Population.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 4.225 (0.518) [lower limit 0.518]
  Week 12 | 3.829 (0.589) [lower limit 0.589]
  Week 24 | 3.515 (1.113) [lower limit 1.113]
  Week 36 | 3.282 (1.263) [lower limit 1.263]
  Week 48 | 3.215 (1.352) [lower limit 1.352]
  FU Week 24 | 3.137 (1.463) [lower limit 1.463]

51. Secondary Outcome: Change From Baseline in Liver Stiffness Measure (LSM) in Groups A, B, C
Description: Liver elastography was performed to assess elasticity and extent of hepatic fibrosis. The change in LSM from Baseline to each visit was averaged among all participants in expressed in kilopascals (kPa). Positive changes in LSM values corresponded to an increase in stiffness and hepatic fibrosis. Liver Substudy Population: All participants who consented to participate in the liver elasticity substudy. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Week 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 44 | 25 | 6
kPa
  Week 48 | -0.49 (2.151) | 0.376 (2.719) | -1.517 (1.685)
  FU Week 24 | -1.026 (2.269) | -0.72 (2.633) | -1.7 (1.033)

52. Secondary Outcome: Percentage of Participants With >15% Drop in Height Percentile for Age in Group C
Description: The percentage of participants with >15% drop in weight percentile for age from Baseline to each visit was reported. Safety Population.
Time Frame: Weeks 30, 36; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Number; unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants
  Week 30 | 20
  Week 36 | 10
  FU Week 4 | 10
  FU Week 12 | 10
  FU Week 24 | 20

53. Secondary Outcome: Change From Baseline in Height for Age Z-Score in Groups A and B
Description: The difference between the population mean and raw scores was calculated as the height for age z-score. Mean absolute values at Baseline were reported. The change from Baseline to each visit was averaged among all participants and expressed in units of standard deviations. Safety Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Weeks 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: standard deviations
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 49
standard deviations
  Baseline | 0.271 (1.149) | -0.062 (1.17)
  Week 12 | 0.011 (0.258) | -0.006 (0.185)
  Week 24 | -0.04 (0.293) | -0.071 (0.264)
  Week 36 | -0.056 (0.337) | -0.025 (0.328)
  Week 48 | -0.099 (0.365) | -0.013 (0.284)
  FU Week 12 | -0.112 (0.404) | -0.037 (0.243)
  FU Week 24 | -0.117 (0.429) | -0.079 (0.282)

54. Secondary Outcome: Change From Baseline in Weight for Age Z-Score in Groups A and B
Description: The difference between the population mean and raw scores was calculated as the weight for age z-score. Mean absolute values at Baseline were reported. The change from Baseline to each visit was averaged among all participants and expressed in units of standard deviations.Safety Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: standard deviations
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 49
standard deviations
  Baseline | 0.106 (1.154) | -0.047 (1.154)
  Week 1: number analyzed (Participants) | 101 | 0
  Week 1 | -0.024 (0.089) |
  Week 2: number analyzed (Participants) | 101 | 0
  Week 2 | -0.023 (0.108) |
  Week 4: number analyzed (Participants) | 101 | 0
  Week 4 | -0.048 (0.158) |
  Week 8: number analyzed (Participants) | 101 | 0
  Week 8 | -0.082 (0.228) |
  Week 12 | -0.09 (0.267) | -0.04 (0.241)
  Week 18: number analyzed (Participants) | 101 | 0
  Week 18 | -0.155 (0.309) |
  Week 24 | -0.165 (0.35) | -0.09 (0.323)
  Week 30: number analyzed (Participants) | 101 | 0
  Week 30 | -0.189 (0.372) |
  Week 36 | -0.192 (0.395) | -0.057 (0.338)
  Week 42: number analyzed (Participants) | 101 | 0
  Week 42 | -0.24 (0.375) |
  Week 48 | -0.214 (0.371) | -0.082 (0.343)
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | -0.156 (0.346) |
  FU Week 12 | -0.089 (0.384) | -0.263 (0.333)
  FU Week 24 | -0.046 (0.452) | -0.322 (0.325)

55. Secondary Outcome: Change From Baseline in Height for Age Z-Score in Group C
Description: The difference between the population mean and raw scores was calculated as the height for age z-score. Mean absolute values at Baseline were reported. The change from Baseline to each visit was averaged among all participants and expressed in units of standard deviations. Safety Population.
Time Frame: Baseline; Weeks 12, 24, 36, 48; FU Weeks 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: standard deviations
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
standard deviations
  Baseline | 0.586 (0.947) [lower limit 0.947]
  Week 12 | 0.07 (0.492) [lower limit 0.492]
  Week 24 | 0.262 (0.42) [lower limit 0.42]
  Week 36 | 0.3 (0.601) [lower limit 0.601]
  Week 48 | 0.19 (0.683) [lower limit 0.683]
  FU Week 12 | 0.205 (0.611) [lower limit 0.611]
  FU Week 24 | 0.064 (0.634) [lower limit 0.634]

56. Secondary Outcome: Change From Baseline in Weight for Age Z-Score in Group C
Description: The difference between the population mean and raw scores was calculated as the weight for age z-score. Mean absolute values at Baseline were reported. The change from Baseline to each visit was averaged among all participants and expressed in units of standard deviations. Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: standard deviations
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
standard deviations
  Baseline | 0.187 (1.141)
  Week 1 | -0.044 (0.052)
  Week 2 | -0.023 (0.107)
  Week 4 | 0.049 (0.243)
  Week 8 | -0.041 (0.198)
  Week 12 | 0.012 (0.288)
  Week 18 | -0.018 (0.377)
  Week 24 | -0.089 (0.245)
  Week 30 | -0.094 (0.34)
  Week 36 | 0 (0.443)
  Week 42 | -0.032 (0.344)
  Week 48 | -0.208 (0.374)
  FU Week 4 | -0.054 (0.35)
  FU Week 12 | -0.156 (0.29)
  FU Week 24 | -0.161 (0.309)

57. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at 24 Weeks After EOT in Group C
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. The percentage of participants with HBeAg seroconversion at 24 weeks after EOT was reported. The 95% CI was calculated by the Pearson-Clopper method. Safety Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
percentage of participants | 30 (6.67) [6.67 to 65.25]

58. Secondary Outcome: Change From Baseline in Quantitative Serum ALT Level in Groups A and B
Description: The change in quantitative ALT from Baseline to each visit was averaged among all participants and expressed as a factor of the laboratory-specific ULN (for example, 1 × ULN, 2 × ULN, 3 × ULN). ITT Population. All participants were included in the endpoint analysis. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: factor of ULN
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
factor of ULN
  Week 1: number analyzed (Participants) | 101 | 0
  Week 1 | 0.606 (1.565) |
  Week 2: number analyzed (Participants) | 101 | 0
  Week 2 | 0.06 (2.283) |
  Week 4: number analyzed (Participants) | 101 | 0
  Week 4 | 0.564 (3.026) |
  Week 8: number analyzed (Participants) | 101 | 0
  Week 8 | 0.463 (3.225) |
  Week 12 | 0.415 (3.732) | 0.598 (5.934)
  Week 18: number analyzed (Participants) | 101 | 0
  Week 18 | 0.288 (3.332) |
  Week 24 | 0.004 (3.496) | -0.462 (2.311)
  Week 30: number analyzed (Participants) | 101 | 0
  Week 30 | -0.1 (3.163) |
  Week 36 | -0.302 (2.8) | -0.51 (1.835)
  Week 42: number analyzed (Participants) | 101 | 0
  Week 42 | -0.436 (2.732) |
  Week 48 | -0.63 (2.652) | -0.939 (1.914)
  FU Week 4: number analyzed (Participants) | 101 | 0
  FU Week 4 | -1.474 (2.889) |
  FU Week 12: number analyzed (Participants) | 101 | 0
  FU Week 12 | -0.736 (2.972) |
  FU Week 24 | -1.302 (2.766) | -0.701 (2.22)

59. Secondary Outcome: Change From Baseline in Quantitative HBeAg Level in Groups A and B
Description: The change in quantitative HBeAg from Baseline to each visit was averaged among all participants and expressed in log10 PEIU/mL. ITT Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 PEIU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 92 | 43
log10 PEIU/mL
  Week 12 | -0.583 (0.672) | -0.225 (0.497)
  Week 24 | -0.834 (0.805) | -0.261 (0.612)
  Week 36 | 1.123 (0.91) | -0.3 (0.621)
  Week 48 | -1.28 (1.043) | -0.491 (0.74)
  FU Week 24 | -1.24 (1.205) | -0.452 (0.793)

60. Secondary Outcome: Change From Baseline in Quantitative HBsAg Level in Groups A and B
Description: The change in quantitative HBsAg from Baseline to each visit was averaged among all participants and expressed in log10 IU/mL. ITT Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 44
log10 IU/mL
  Week 12 | -0.444 (1.021) | -0.081 (0.356)
  Week 24 | -0.798 (1.343) | -0.032 (0.392)
  Week 36 | -1.051 (1.534) | -0.126 (0.26)
  Week 48 | -1.239 (1.652) | -0.188 (0.285)
  FU Week 24 | -0.936 (1.491) | -0.204 (0.316)

61. Secondary Outcome: Change From Baseline in Quantitative Serum ALT Level in Group C
Description: The change in quantitative ALT from Baseline to each visit was averaged among all participants and expressed as a factor of the laboratory-specific ULN (for example, 1 × ULN, 2 × ULN, 3 × ULN). Safety Population. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48; FU Weeks 4, 12, 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: factor of ULN
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
factor of ULN
  Week 1 | 0.313 (0.414)
  Week 2 | 0.091 (0.991)
  Week 4 | -0.361 (1.566)
  Week 8 | -0.101 (1.895)
  Week 12 | -0.012 (1.613)
  Week 18 | -0.589 (0.996)
  Week 24 | -0.917 (1.31)
  Week 30 | -0.584 (1.73)
  Week 36 | -0.633 (1.455)
  Week 42 | -1.211 (1.05)
  Week 48 | -1.104 (1.084)
  FU Week 4 | -1.669 (0.95)
  FU Week 12 | -1.283 (1.501)
  FU Week 24 | -1.256 (1.757)

62. Secondary Outcome: Change From Baseline in Quantitative HBeAg Level in Group C
Description: The change in quantitative HBeAg from Baseline to each visit was averaged among all participants and expressed in log10 PEIU/mL. Safety Population. "Number of subjects analyzed" reflects the total number of participants who provided evaluable data at any timepoint. The number of participants who provided evaluable data for the analysis at each timepoint (n) is shown in the table.
Time Frame: Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 PEIU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 PEIU/mL
  Week 12 | -0.779 (0.645)
  Week 24 | -0.817 (0.678)
  Week 36 | -0.817 (0.685)
  Week 48 | -0.762 (0.818)
  FU Week 24 | -0.742 (0.84)

63. Secondary Outcome: Change From Baseline in Quantitative HBsAg Level in Group C
Description: The change in quantitative HBsAg from Baseline to each visit was averaged among all participants and expressed in log10 IU/mL. Safety Population.
Time Frame: Weeks 12, 24, 36, 48; FU Week 24 (up to 72 weeks overall)
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group C: PEG-IFN Monotherapy With Advanced Fibrosis
Number analyzed (Participants) | 10
log10 IU/mL
  Week 12 | -0.397 (0.428) [lower limit 0.428]
  Week 24 | -0.71 (0.712) [lower limit 0.712]
  Week 36 | -0.943 (0.913) [lower limit 0.913]
  Week 48 | -1.01 (1.019) [lower limit 1.019]
  FU Week 24 | -1.088 (1.141) [lower limit 1.141]

64. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion Over Time in Groups A and B
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: Baseline, FU Years: 1, 2, 3, 4, 5
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis
Number analyzed (Participants) | 101 | 50
percentage of subjects
  Baseline | 0.00 (0.00) [0.00 to 3.59] | 0.00 (0.00) [0.00 to 7.11]
  Fu Year 1 | 32.7 (23.67) [23.67 to 42.72] | 6.08 (1.25) [1.25 to 16.55]
  Fu Year 2 | 33.7 (24.56) [24.56 to 43.75] | 6.08 (1.25) [1.25 to 16.55]
  Fu Year 3 | 46.5 (36.55) [36.55 to 56.73] | 6.08 (1.25) [1.25 to 16.55]
  Fu Year 4 | 30.7 (21.90) [21.90 to 40.66] | 8.00 (2.22) [2.22 to 19.23]
  Fu Year 5 | 5.9 (2.21) [2.21 to 12.48] | 0.00 (0.00) [0.00 to 7.11]

65. Secondary Outcome: Percentage of Participants With Loss of HBeAg at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 2
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group D: Switch to PEG-IFN Monotherapy: Participants without advanced fibrosis who did not receive treatment and had not experienced HBeAg seroconversion were allowed to switch to PEG-IFN monotherapy: 4.5-year extended follow-up
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 30.3 [15.59 to 48.71]

66. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 1
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 9.1 [1.92 to 24.33]

67. Secondary Outcome: Percentage of Participants With Loss of HBsAg at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 1
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 12.1 [3.40 to 28.20]

68. Secondary Outcome: Percentage of Participants With Normal ALT at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 13
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 42.4 [25.48 to 60.78]

69. Secondary Outcome: Percentage of Participants With HBV Deoxyribonucleic Acid (DNA) <20,000 International Units Per Milliliter (IU/mL) at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 5
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 36.4 [20.40 to 54.88]

70. Secondary Outcome: Percentage of Participants With HBV DNA <2,000 IU/mL at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 6
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 27.3 [13.30 to 45.52]

71. Secondary Outcome: Percentage of Participants With HBV DNA Undetectable at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: HBV DNA was quantified using PCR by Roche Taqman. Undetectable HBV DNA was defined as HBV DNA <29 IU/mL. The percentage of participants with HBV DNA undetectable at 24 weeks after EOT/POP was reported. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 18.2 [6.98 to 35.46]

72. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <20,000 IU/mL at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: HBeAg seroconversion was defined as loss of HBeAg and the presence of anti-HBe. HBV DNA was quantified using PCR by Roche Taqman. The 95% CI was calculated by the Pearson-Clopper method. ITT Population.
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 27.3 [13.30 to 45.52]

73. Secondary Outcome: Percentage of Participants With Combined HBeAg Seroconversion and HBV DNA <2,000 IU/mL at 24 Weeks After the End of Switch Treatment Period: Switch Group
Description: as for outcome 8
Time Frame: FU Week 24 (up to 72 weeks overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group D: Switch to PEG-IFN Monotherapy
Number analyzed (Participants) | 33
percentage of participants | 21.2 [8.98 to 38.91]

ADVERSE EVENTS:
Time Frame: From Baseline to approximately 4.5 years
Description: Safety Population
Groups:
- Group A: PEG-IFN Monotherapy Without Advanced Fibrosis: Participants without advanced fibrosis were randomized and received PEG-IFN monotherapy for 48 weeks with a 24-week follow-up and an additional ongoing 4.5-year extended follow-up. Each dose of 45 to 180 mcg was based on BSA and given as a once-weekly SC injection for 48 weeks. BSA-based dosing was as follows: 0.51-0.53 m^2, 45 mcg; 0.54-0.74 m^2, 65 mcg; 0.75-1.08 m^2, 90 mcg; 1.09-1.51 m^2, 135 mcg; >1.51 m^2, 180 mcg.
- Group B: Untreated Control Without Advanced Fibrosis: Participants without advanced fibrosis were randomized and were evaluated for 48 weeks with a 24-week follow-up and an additional ongoing 4.5-year extended follow-up. As the study is open-label, participants did not receive any investigational or placebo treatment during the 48-week POP. For ethical reasons, participants in Group B had a reduced visit schedule (every 12 weeks) compared to participants in Group A through the end of 24-week follow-up.
- Group C: PEG-IFN Monotherapy With Advanced Fibrosis: Participants with advanced fibrosis were allocated (not randomized) to receive PEG-IFN monotherapy for 48 weeks with a 24-week follow-up and an additional ongoing 4.5-year extended follow-up. Each dose of 45 to 180 mcg was based on BSA and given as a once-weekly SC injection for 48 weeks. BSA-based dosing was as follows: 0.51-0.53 m^2, 45 mcg; 0.54-0.74 m^2, 65 mcg; 0.75-1.08 m^2, 90 mcg; 1.09-1.51 m^2, 135 mcg; >1.51 m^2, 180 mcg.
- Group A - Long Term Follow-up; Group B - Long Term Follow-up: Participants without advanced fibrosis: 4.5-year extended follow-up
- Group C Long Term Follow-up: Participants with advanced fibrosis: 4.5-year extended follow-up
- Group D - Long Term Follow-up: Participants without advanced fibrosis who did not receive treatment and had not experienced HBeAg seroconversion were allowed to switch to PEG-IFN monotherapy: 4.5-year extended follow-up
Arm/Group | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis | Group B: Untreated Control Without Advanced Fibrosis | Group C: PEG-IFN Monotherapy With Advanced Fibrosis | Group D: Switch to PEG-IFN Monotherapy | Group A - Long Term Follow-up | Group B - Long Term Follow-up | Group C Long Term Follow-up | Group D - Long Term Follow-up
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/49 | 0/10 | 0/33 | 0/101 | 0/49 | 0/10 | 0/33
Serious Adverse Events (participants affected / at risk) | 6/101 | 1/49 | 0/10 | 2/33 | 0/101 | 0/49 | 0/10 | 0/33
Other Adverse Events (participants affected / at risk) | 80/101 | 18/49 | 9/10 | 21/33 | 25/101 | 6/49 | 0/10 | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis (N=101) | Group B: Untreated Control Without Advanced Fibrosis (N=49) | Group C: PEG-IFN Monotherapy With Advanced Fibrosis (N=10) | Group D: Switch to PEG-IFN Monotherapy (N=33) | Group A - Long Term Follow-up (N=101) | Group B - Long Term Follow-up (N=49) | Group C Long Term Follow-up (N=10) | Group D - Long Term Follow-up (N=33)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microsporum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: PEG-IFN Monotherapy Without Advanced Fibrosis (N=101) | Group B: Untreated Control Without Advanced Fibrosis (N=49) | Group C: PEG-IFN Monotherapy With Advanced Fibrosis (N=10) | Group D: Switch to PEG-IFN Monotherapy (N=33) | Group A - Long Term Follow-up (N=101) | Group B - Long Term Follow-up (N=49) | Group C Long Term Follow-up (N=10) | Group D - Long Term Follow-up (N=33)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 10 (26) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 10 (10)
Fatigue (General disorders) | 9 (12) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Influenza like illness (General disorders) | 15 (18) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 49 (107) | 5 (8) | 8 (14) | 17 (35) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 5 (8) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (10) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 9 (10) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Body temperature increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (20) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 30 (71) | 2 (2) | 4 (9) | 11 (14) | 1 (1) | 0 (0) | 0 (0) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 19 (30) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (10) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (16) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (9) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (14) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (17) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (14) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingiviti (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticardia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase mb increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B DNA increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duane's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Accommodation disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Expired product administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-05-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT01519960/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT01519960/SAP_001.pdf